CLINICAL TRIAL: NCT06928649
Title: Innovative Cell Death Diagnostics Allowing Stratifying Critically Ill Patients for Novel Ferroptosis or Pyroptosis Intervention Strategies
Brief Title: Stratifying Critically Ill Patients for Novel Ferroptosis or Pyroptosis Intervention Strategies
Acronym: ICU-FERRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Philppe Jorens, Prof., University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDGE 3060
Record Dates: First submitted 2025-03-24; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Trauma Related Injuries; Subarachnoid Haemorrhage (SAH)
MeSH Terms: conditions — Sepsis; Subarachnoid Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Critical illness (Experimental): Patient who are admitted to the ICU, with a predicted length of stay > 48 hours. Admission due to sepsis, trauma, haemorrhagic shock, neurological catastrophe
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood sampling: 3 first days of admision, 2 ml of plasma daily Urine, BALF, CSF sampling: 1 day during 3 first days of admission
  Other Names: Urine sampling; Bronchoalveolar lavage sampling; Cerebrospinal fluid sampling

SUMMARY:
In order to better determine which therapy is best for patiënts which present with organ falure during the course of their stay in the intesive care unit (ICU) , one has to determine which underlying mechanism is causing this organ falure. We will determine levels of so called "biomarkers" for ferroptosis (a mechan ism of iron-related cell death) in the peripheral blood and biological fluids of criticaly ill patients admitted to the ICU with a catastrrophy (severe infection, trauma ...) . Why ? If it turns out that this ferroptosis plays a role in the ocurrence of organ failure in the critially ill, this will lead to new therapies in the future as drugs become more and more available which can influene this biochemical "pahway". of iron-relatd death.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU of UZA
* Critically ill and predicted to be hospitalised in the ICU for > 48 hours (i.e. mostly patients admitted for sepsis, trauma, haemorrhagic shock, neurological catastrophe … which means at risk to develop mono-or multiple organ failure)
* With arterial line in place (for blood sampling)

Exclusion Criteria:

* Refusal of consent by patient or closest relative
* Postoperative patients after major surgery in whom prolonged ICU stay is not foreseen (i.e. elective cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with survival after 28 days. | 28 days
  Survival in and after ICU.

SECONDARY OUTCOMES:
Change from baseline concentration of Norepinephrine every day during ICU stay | 28 days
Change in SOFA score during ICU stay | Change from enrollment to 14 days of ICU stay
  SOFA score, with a higher score for more severe organ failure

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jorens, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Undecided